CLINICAL TRIAL: NCT04426773
Title: Electroencephalography (EEG) Predictors of Response to Transcranial Direct Current Stimulation (tDCS) Treating Obsessive-Compulsive Disorder (OCD)
Brief Title: Electroencephalography (EEG) Predictors of Transcranial Direct Current Stimulation (tDCS) in Obsessive-Compulsive Disorder (OCD)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai Mental Health Center (Other)
Responsible Party: Principal Investigator, Zhen Wang, vice-president, Shanghai Mental Health Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SMHC-OCD-006
Record Dates: First submitted 2020-06-08; First posted 2020-06-11 (Actual); Last update posted 2025-05-15 (Actual); Status verified 2025-05

CONDITIONS: Obsessive-Compulsive Disorder
Keywords: transcranial direct current stimulation
MeSH Terms: conditions — Obsessive-Compulsive Disorder

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- tDCS treatment (Experimental): Cathode transcranial direct current stimulation over the right OFC will be applied once a day, 5 days a week, for 2 weeks.
  Interventions: Device: High-Definition transcranial direct current stimulation

INTERVENTIONS:
Device: High-Definition transcranial direct current stimulation — The tDCS device will deliver a direct current of 1.5mA for 20 minutes. Cathode electrode will be localized in front of the OFC on the Fp2 point according to the EEG international reference. Four anode electrodes will be placed around FP2 (i.e. Fpz, AFz, AF4, AF8).

SUMMARY:
This study is designed to find Electroencephalogram (EEG) biomarkers to predict transcranial direct current stimulation (tDCS) response in obsessive-compulsive disorder.

DETAILED DESCRIPTION:
The purpose of this study is to explore resting state electroencephalography and transcranial magnetic stimulation and electroencephalography (TMS-EEG) biomarkers that would predict transcranial direct current stimulation (tDCS) response in obsessive-compulsive disorder with cathode electrode targeting orbitofrontal cortex (OFC). 30 OCD patients will be recruited to this study and performed once a day, five times a week direct current stimulation treatment for two weeks. The investigators will assess symptom severity before and after two weeks of tDCS. Through the study, Yale-Brown Obsessive Compulsive Scale（Y-BOCS）, the Obsessive Compulsive Inventory-Revised (OCI-R), the Beck Depression Inventory(BDI), Pittsburgh sleep quality index (PSQI)and side-effect questionnaire will be obtained by a trained investigator. Resting state electroencephalography and TMS-EEG testing will be conducted before and after tDCS treatment.

ELIGIBILITY:
Inclusion Criteria:

* age: 18-50 years old;
* DSM-5 criteria for OCD;
* Y-BOCS total score > or = 16
* >or＝9 years education

Exclusion Criteria:

* any additional current psychiatric comorbidity
* The inability to receive tDCS because of metallic implants, or history of seizures，history of head injury, or history of neurosurgery.
* Participants with claustrophobic, heart pacemaker, mechanical heart valve, mechanical implant such as an aneurysm clip, hip replacement, or any other pieces of metal that have accidentally entered their body.
* Any current significant medical condition.
* serious suicide risk

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2020-07-01 (Actual); Primary Completion 2025-04-30 (Actual); Study Completion 2025-05-01 (Actual)

PRIMARY OUTCOMES:
Change in symptom improvement assessed by the Yale-Brown Obsessive Compulsive Scale (Y-BOCS) | Up to 3 months
  It assesses the severity of OCD symptoms. The Y-BOCS scale ranges from 0 to 40, with 0 being no symptoms and 40 being severe.The responder on Y-BOCS is defined as a Y-BOCS decrease at least 35% from the baseline at post-treatment.
Change in long-interval intracortical inhibition (LICI) and short interval intracortical inhibition (SICI) measured by TMS-EEG | Up to 2 weeks
  LICI and SICI are TMS-EEG paradigm to assess the extent of cortical inhibition. LICI and SICI will be measured using single and paired TMS pulses applied to the OFC. LICI and SICI will be compared between before and after treatment.
EEG biomarkers as predictors of response to tDCS | baseline
  LICI and SICI measured by TMS-EEG and resting state EEG will be performed to investigate predictors of response to tDCS in OCD patients.

SECONDARY OUTCOMES:
Change in Obsessive Compulsive Inventory-Revised(OCI-R) | Up to 3 months
  It is an inventory of OCD symptoms with 18 items that are rated on a 5-point Likert scale. Total scores range from 0 to 72, with higher scores indicating more severe OCD symptoms.
Change in The Beck Depression Inventory(BDI) | Up to 3 months
  It consists of 21 items and uses a 0 to 3 severity scale. Total scores range from 0 to 63, with higher scores indicating more severe depression symptoms.
Change in The Beck Anxiety Inventory (BAI) | Up to 3 months
  It is an inventory of anxiety symptoms with 18 items that are rated on a 5-point Likert scale(0 to 4). Total scores range from 0 to 72, with higher scores indicating more severe anxiety symptoms.
Change in Pittsburgh sleep quality index(PSQI) | Up to 3 months
  The Pittsburgh Sleep Quality Index (PSQI) contains 19 self-rated questions which measures seven aspects of sleep: (1) subjective sleep quality, (2) sleep latency, (3) sleep duration, (4) habitual sleep efficiency, (5) sleep disturbances, (6) use of sleeping medication, and (7) daytime dysfunction. The 19 self-rated items are combined to form seven component scores, each of which has a range of 0-3 points (0 indicates no difficulty, while 3 indicates severe difficulty). The seven component scores are then summed to yield one global score, with a range of 0-21 points (0 indicating no difficulty, and 21 indicating severe difficulties in all the seven areas of sleep quality).
Change in Side-effect questionnaire | Up to 3 months
  It consists of 10-item and uses 0 to 3 severity scale to rate the intensity of side effects. Total scores range from 0 to 30, with higher scores indicating more severe side-effect. It also assesses the relation between side-effect and the effects of tDCS using 0 to 4 scale. Total scores range from 0 to 40, with higher score indicating the greater relation.

CONTACTS AND LOCATIONS:
Overall Officials: Zhen Wang, PhD,MD, Principal Investigator — Shanghai Mental Health Center
Locations (1):
- Shanghai Mental Health Center, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No